CLINICAL TRIAL: NCT05987189
Title: Diagnostic Performance of Small RNA Blood Test in Patients Undergoing Follow-up Imaging After Positive Low Dose CT Screening for Cancer of the Lung "Early Detection of Lung Cancer Based on Small RNA Signatures - Boston II"
Brief Title: Diagnostic Performance of Small RNA Blood Test in Patients Undergoing Follow-up Imaging After Positive Low Dose CT Screening for Cancer of the Lung
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hummingbird Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: Boston II
Record Dates: First submitted 2023-04-26; First posted 2023-08-14 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — *Blood sample (2x2,5 ml blood in PAXgene® tubes, 1x10 ml Streck® RNA Complete BCT CE blood, 1x10 ml Streck® Cell-free DNA BCT CE blood)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: miLungDx — At study enrollment a blood sample will be drawn prior to any invasive diagnostic study or treatment. On this blood sample a novel lung cancer test relying on small RNA signatures will be performed and evaluated.

SUMMARY:
2,000 individuals, aged 50-80 who have received a lung-RADS category 3 or 4 result on a LDCT screening study and who are scheduled for follow-up diagnostic imaging study, biopsy, clinical consultation or surgical appointment at one of the participating hospitals.

DETAILED DESCRIPTION:
The study is a prospective, longitudinal, observational study to evaluate the performance of a novel diagnostic test for early-stage lung cancer.

Study duration: Expected patient enrollment to be completed within 12 months after study initiation. Patients will be followed for a minimum of 12 months from the date of enrollment. The study duration is approximately 2 years.

Participant duration: The day of blood collection. Participants will follow their regular standard of care schedule as recommended by existing guidelines; no extra visits are planned. Follow up data will be obtained from the electronic medical record within at least 12 months of follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients, aged 50 to 80 years
* Received a lung RADS category 3 or 4 finding on a LDCT screening exam (first or subsequent) and are referred to undergo further diagnostic procedures for the detection of lung cancer
* Has undergone LD-CT screening exam within last 90 days and allows for blood sampling within this period
* Subject may not have undergone any invasive diagnostic procedure in relation to the suspicious nodule
* Able and willing to provide informed consent

Exclusion Criteria:

* Prior history of diagnosed lung cancer
* History of gastrointestinal, hematological, breast, thyroid, and genitourinary cancer within the past 10 years
* Active infectious diseases, such blood borne viral diseases (e.g. AIDS, hepatitis)
* Immunosuppressive medication
* Deemed not able to participate in the study by the investigator

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals, aged 50-80 who have received a lung-RADS category 3 or 4 result on a LDCT screening study and who are scheduled for follow-up diagnostic imaging study, biopsy, clinical consultation or surgical appointment at one of the participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 1 year
  The study is a prospective, longitudinal, observational study to evaluate the performance of a novel diagnostic test for early-stage lung cancer. The primary endpoint is to detect the presence or absence of lung cancer, as determined by all follow-up imaging, and pathological data obtained throughout the duration of the study.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Northside Hospital, Atlanta, Georgia
  - Mass General Brigham, Boston, Massachusetts
  - Henry Ford Health, Detroit, Michigan
  - Jacobi Medical Center, The Bronx, New York
  - New York Health + Hospitals, The Bronx, New York
  - Duke University Health System, Durham, North Carolina
  - Baptist Hospitals of Southeast Texas, Beaumont, Texas
  - University Of Utah Health, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No